CLINICAL TRIAL: NCT01382784
Title: Psoriasis and the Risk of Cardiovascular Disease. A Prospective Observational Study to Detect Cardiovascular Risk Factors
Brief Title: Psoriasis and the Risk of Cardiovascular Disease. A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Responsible Party: Ellen Slevolden, medical doctor, department of Dermatology, Oslo university Hospital
Other Study IDs: Psoriasis and comorbidity
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-05

CONDITIONS: Psoriasis; Cardiovascular Disease
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is growing evidence that psoriasis is a systemic disorder which enhances atherosclerosis and the risk of cardiovascular disease. Epidemiological studies have shown an independent association between psoriasis and atherosclerosis, stroke and coronary artery disease. The main goal of this on-going study is to register data which will enable the identification of new markers of atherosclerosis activity and carotid plaque instability in patients with severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old, psoriasis for more than 5 years, moderate to severe psoriasis (PASI >10 or systemic treatment)

Exclusion Criteria:

* familiar hypercholesterolemia, ongoing infections and cancer disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have had psoriasis for more than 5 years are being admitted to the study. The assessments include: clinical data, treatment, platelet aggregation and blood viscosity, serum markers and mediators of atherosclerosis, carotid IMT and plaque burden assessed by Color Duplex ultrasound. The patients are recruited from our dermatological department (in and outdoor patients)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-05

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Dermatological Department, OUS, Oslo
  - Oslo university Hospital, Dermatological dept, Oslo